CLINICAL TRIAL: NCT04201860
Title: Blood Gas and Bleeding Disorders in Healthy Volunteers Exposed to Nitroglycerin and Nitrogen Compounds of Blasting Gelatin: a Field Report During a Cave Accident
Brief Title: Blood Gas and Bleeding Disorders in Healthy Volunteers Exposed to Nitroglycerin and Nitrogen Compounds
Status: Completed | Type: Observational
Sponsor: Emiliano Petrucci (Other)
Responsible Party: Sponsor-Investigator, Emiliano Petrucci, Principal Investigator, San Salvatore Hospital of L'Aquila
Organization: San Salvatore Hospital of L'Aquila (Other)
Other Study IDs: 20/2016
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Disorder of Blood Gas; Bleeding Disorder
Keywords: Arterial blood gas; Coagulation; Nitrogen compounds
MeSH Terms: conditions — Hemostatic Disorders; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Blasters group: The volunteers of the blasters group of Italian Mountain and Cave Rescue handled explosive with nitrogen compounds and nitroglycerin of micro-charges, before the accidental uncontrolled detonation.
  Interventions: Diagnostic Test: Arterial blood gas analyses and haemostasis measures
- Not blasters group: The volunteers of the blasters group of Italian Mountain and Cave Rescue did not handle explosive with nitrogen compounds and nitroglycerin of micro-charges, before the accidental uncontrolled detonation.
  Interventions: Diagnostic Test: Arterial blood gas analyses and haemostasis measures

INTERVENTIONS:
Diagnostic Test: Arterial blood gas analyses and haemostasis measures — Under aseptic conditions, a puncture of radial artery was performed: three mL of the arterial blood sample were used for the haemostasis measure, while one mL was tested for the blood gases analysis.

SUMMARY:
The aim of the study was to investigate the possible relationship about blood gas and bleeding disorders in healthy volunteers of blasters and no blasters groups of the Italian National Mountain and Cave Rescue who handled nitrogen compounds and nitroglycerine and then they were exposed to combustion products from an accidental uncontrolled detonation of micro-charges during a cave unblocking procedure.

DETAILED DESCRIPTION:
This was a field report of clinical data collected during an accidental uncontrolled detonation of micro-charges, while the cave unblocking procedure was performed by volunteers of blaster group and non blasters group of the Italian National Mountain and Cave Rescue, in a cave in Trieste (Italy; altitude entrance: 348 meters above sea level; total length: 413,5 meters; total depth of 307 meters).

Before going into the cave (Time 0), the following clinical data were collected: age, sex, body mass index; smoke (yes/no), heart rate, arterial blood pressure (mean arterial pressure), oxygen saturation measured with pulse oxymetry, epitympanic temperature, blood gases analyses and the haemostasis measures.

After the accidental uncontrolled detonation of micro-charges, (Time 1) heart rate, arterial blood pressure, oxygen saturation measured with pulse oxymetry, epitympanic temperature, blood gases analyses and the haemostasis measures were recorded in each volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of Italian National Mountain and Cave Rescue

Exclusion Criteria:

* gas exchange disorders
* quantitative abnormalities of coagulation assessment
* qualitative abnormalities of coagulation assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers of Blasters and No Blasters Group of the Italian National Mountain and Cave Rescue
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline arterial blood gases analysis at 2 hours | 10 minutes before going in to the cave and two hours after the volunteers come out from the cave
  Under aseptic conditions, a puncture of radial artery was performed: one mL was tested for the blood gases analysis, by using i-STAT analyser.
Change from baseline haemostasis analysis at 2 hours | 10 minutes before going in to the cave and two hours after the volunteers come out from the cave
  Under aseptic conditions, a venipuncture was performed: three mL of blood sample were used for the haemostasis measure, by using Rotational Thromboelastometry

SECONDARY OUTCOMES:
Change from Baseline heart rate at 2 hours | 10 minutes before going in to the cave and two hours after the volunteers come out from the cave
  Haert rate was recorded by using a multiparametric monitor
Change from baseline arterial blood pressure at 2 hours | 10 minutes before going in to the cave and two hours after the volunteers come out from the cave
  Arterial blood pressure was recorded by using a multiparametric monitor
Change from baseline pulse oxymetry at 2 hours | 10 minutes before going in to the cave and two hours after the volunteers come out from the cave
  Pulse oxymetry was recorded by using a multiparametric monitor
Change from baseline epitympanic temperature at 2 hours | 10 minutes before going in to the cave and two hours after the volunteers come out from the cave
  Epitympanic temperature was measured by using epitympanic probe

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Petrucci, MD, Study Chair — San Salvatore Academic Hospital
Locations (1):
- Barbara Pizzi, Avezzano, Italy

IPD SHARING:
Plan to Share IPD: No